CLINICAL TRIAL: NCT03750214
Title: Bio Colposcopy System CIP: Evaluation of the Biop Colposcopy System's Safety and Performance (Accuracy of Its Registration Procedure)
Brief Title: Evaluation of the Biop Colposcopy System's Safety and Performance (Accuracy of Its Registration Procedure)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BIOP Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLP - 430
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biop Coplposcopy System (Experimental): Biop Colposcopy system procedure
  Interventions: Device: Biop Colposcopy System

INTERVENTIONS:
Device: Biop Colposcopy System — The procedure stages:
  1. Scanning of the cervix - the cervix is scanned using the micro colposcope probe unit, to produce a total of 51 micro-images and one macro image from the panoramic camera.
  2. Colposcopy exam - during the standard colposcopy exam, the doctor acquires a panoramic image of the cervix with the digital colposcope.
  3. A questionnaire completed by the subject after the Biop procedure, with regards to any unusual sensations or events experienced during the procedure.
  4. A questionnaire completed by the user after the Biop procedure, with regards to system usage
  5. Image Registration analysis

SUMMARY:
This is a multi-center, prospective, non-randomized, confirmatory study to evaluate the safety and performance of the Biop Digital Colposcope and the accuracy of the image registration procedure between the Biop Digital Colposcope unit and the Biop Micro Colposcope probe unit.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-randomized, confirmatory study to evaluate the safety and performance of the Biop Digital Colposcope and the accuracy of the image registration procedure between the Biop Digital Colposcope unit and the Biop Micro Colposcope probe unit.

The Biop Digital Colposcope is intended for magnified viewing of the tissues of the vagina, cervix and external genitalia in order to assist doctors in diagnosing abnormalities such as lesions or cancer, and selecting areas for biopsy. The images from the digital colposcope are to be viewed on a color display. The digital colposcope is intended for use in hospitals, clinics, and doctor's offices.

The Biop Micro Colposcope probe unit is an imaging tool intended to be placed in the vagina for acquisition of images of the cervix. It is intended as an adjunct to the Biop Digital Colposcope. It should NOT be used as a substitute for a thorough colposcopic evaluation. The Biop Micro Colposcope Probe unit is not intended for use on the vulva and vagina.

It is anticipated that it will take approximately 3 months to complete active enrollment. Study duration for each subject is 1-2 days, including screening, enrolment and procedure. The study will be completed when the final study subject has completed the procedure.

1. Performance - to confirm that average image registration error is less than or equal to (≤) 2mm.
2. Safety - to evaluate the safety of the Biop Digital Colposcope in women undergoing cervical colposcopy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Females, ages 22 to 65 years old
* Referred for colposcopy, following abnormal cervical cytology
* Subject provides signed informed consent

Exclusion Criteria:

* Currently pregnant or nursing
* Currently menstruating
* Currently has intrauterine device (IUD)
* Diagnosed with diseases that may influence the color of the tissue, e.g., hepatitis, polycytemia vera.
* Diagnosed with pathologies that affect blood coagulation, the immune system or undergoing any treatment that interfere with coagulation or the immune system
* HIV-positive status
* Psychological instability, inappropriate attitude or motivation
* Use of any additional experimental drug or device or participation in another clinical study within the past 30 days

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, ages 22 to 65 years old
Enrollment: 26 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Performance | procedure day ± 1 day
  The primary performance endpoint is the image registration success. Image registration success is defined by the registration error (distance between corresponding control points following registration). Average image registration error should be less than or equal to (≤) to 2mm.
frequency and incidence of all Adverse Events | procedure day ± 1 day
  Safety endpoints include frequency and incidence of all Adverse Events (AE) and Serious Adverse Events (SAE) related and unrelated to the device use.

OTHER OUTCOMES:
Exploratory Endpoint | procedure day ± 1 day
  Subject's comfort - as measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ram Eitan, Md., Principal Investigator — RMC Israel

IPD SHARING:
Plan to Share IPD: No